CLINICAL TRIAL: NCT03860025
Title: "Patient Reported Outcome After Dislocation of a Primary THA"
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 3-3013-2128/2
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Quality of Life; Hip Dislocation
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Single dislocation.: Patients with a single postoperative hip dislocation without subsequent revision surgery.
  Interventions: Other: No intervention.
- Recurrent dislocation.: Patients with two or more postoperative hip dislocations without subsequent revision surgery.
  Interventions: Other: No intervention.
- Revision due to dislocation.: Patients with one or more postoperative hip dislocations with subsequent revision surgery due to recurrent instability.
  Interventions: Other: No intervention.
- Controls.: Matched patients without postoperative hip dislocation or revision of any reason.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — No intervention.

SUMMARY:
The aim is to compare QOL and hip specific outcome measures in patients with a single or recurrent episode(s) of THA dislocation and patients with a THA without any dislocation.

DETAILED DESCRIPTION:
Knowledge about the patient's own perception of both general health and more hip-related issues after experiencing a hip dislocation is lacking (19). Hip surgeons need this information in order to incorporate it with other objective aspects, when advising patients with their first hip dislocation. Due to the large study population, this study will provide solid information of what to expect after a hip dislocation and be the largest study ever conducted within this topic. Depending on the results, this study may change the path we choose to advise for our patients after single or recurrent dislocations.

A matched case-control study involving the share of THA patients with at least 1 episode of hip dislocation.

The patients had undergone primary surgery in the 5-year period from 01.01.2010 - 31.12.2014 and subsequent dislocation was evaluated in a 2-year follow-up period. Given a 3-5% approximated incidence of dislocation, 1100-1800 cases will have been identified.

Patients are subdivided in groups depending on the number of dislocations and one group containing THA revisions. In order to be included, a time frame of at least 0,5 year since the last episode of dislocation or surgery must have passed.

A matched control group of patients with primary THA without any event of dislocation are located from the original 5-year period of primary surgery. They will be matched with the group of patients with dislocation, regarding to:

1. Age (+/- 5 years)
2. Gender
3. Date of surgery and hospital

The study will be conducted in accordance with the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guidelines.

After 01.01.2019, all patients included will be receiving 3 questionnaires (a generic - EQ-5D, a hip-specific - HOOS, and an activity scale - UCLA) by e-boks (a mandatory secure email system couplet to the patient's CPR number). Some elderly are exempt and will instead receive the questionnaires by regular mail and a pre-labeled return envelope is attached. Reminders are sent after 2 months.

ELIGIBILITY:
Inclusion Criteria:

* patients with one or more events of hip dislocation after a primary THA
* controls with a primary THA without events of hip dislocation

Exclusion Criteria:

-

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients had undergone primary surgery in the 5-year period from 01.01.2010 - 31.12.2014 and subsequent dislocation was evaluated in a 2-year follow-up period. Cases are found in a previously described study (Protocol-ID 3-3013-2128/1). 1100-1800 cases will be identified, anticipated.
  A matched control group of patients with primary THA without any event of dislocation are located from the original 5-year period of primary surgery. They will be matched with the group of patients with dislocation, regarding to:
  1. Age (+/- 5 years)
  2. Gender
  3. Date of surgery and hospital
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
QOL (Quality of life) | 9 years
  Measured by the EQ-5D questionnaire.
Hip function | 9 years
  Measured by the HOOS questionnaire.

SECONDARY OUTCOMES:
Activity | 9 years
  Measured by the UCLA activity questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lars L. Hermansen, MD, Principal Investigator — Department of Clinical Research, Odense University Hospital, Odense, Denmark.
Locations (1):
- Hospital of South West Jutland, Esbjerg, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Data not to be shared.